CLINICAL TRIAL: NCT01419847
Title: A Prospective, Double-blind, Placebo-controlled Trial of Topical Penlac Nail Lacquer for Therapy of Onychomycosis in Children
Brief Title: Topical Penlac Nail Lacquer for Onychomycosis in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rady Children's Hospital, San Diego (Other)
Responsible Party: Sheila F. Frieldander, MD; PI, Rady Children's Hopsital, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02082C (10856)
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2006-05

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — Ciclopirox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- topical Penlac nail lacquer (Active Comparator): 3-1 randomization of active to placebo
  Interventions: Drug: Ciclopirox
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclopirox
  Arms: topical Penlac nail lacquer
Drug: Placebo
  Arms: Placebo

SUMMARY:
Five months of therapy is sufficient to treat onychomycosis in children. Topical therapy of onychomycosis in children with Penlac nail lacquer has comparable efficacy and a superior cost and safety profile compared to systemic therapy.

DETAILED DESCRIPTION:
Therapeutic trials for the treatment of onychomycosis have been conducted in the adult population, but there is limited data available in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of two and sixteen years
* Clinical diagnosis of toenail onychomycosis involving at least 20% of one nail plate
* Positive DTM reading or fungal culture for onychomycosis-either dermatophytes or non-dermatophyte mold
* Consent to participate in the study
* Women of child-bearing potential must have a negative urine pregnancy test at the baseline visit and be willing to practice effective contraception for the duration of the study.

Exclusion Criteria:

* Children with allergy to Penlac or one of its ingredients
* Structural deformity of target nail plate
* Presence of active psoriasis or severe foot eczema
* Presence of immunodeficiency disorder
* Concurrent immune suppressive therapy or immune suppressive therapy within the last 3 months
* Previous systemic antifungal therapy within the last 6 months
* Previous topical antifungal therapy within the last 14 days
* Female subjects who are pregnant, nursing mothers, those planning a pregnancy during the course of the study, or who become pregnant

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2002-03; Primary Completion 2005-12 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Mycological cure or global evaluation of 2 or less Mycological Cure | Week 20

SECONDARY OUTCOMES:
Estimated cost of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Sheila F Friedlander, MD, Principal Investigator — Rady Children's Hospital, San Diego
Locations (1):
- Children's Hospital-San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Friedlander SF, Chan YC, Chan YH, Eichenfield LF. Onychomycosis does not always require systemic treatment for cure: a trial using topical therapy. Pediatr Dermatol. 2013 May-Jun;30(3):316-22. doi: 10.1111/pde.12064. Epub 2012 Dec 28. PMID 23278851